CLINICAL TRIAL: NCT05003232
Title: NIRS Directed Optimal Cerebral Perfusion Pressure on the Outcome of Aneurysmal Subarachnoid Hemorrhage Patients: A Multicenter, Single-blinded, Randomized Controlled Trial
Brief Title: NIRS Directed Optimal Cerebral Perfusion Pressure on the Outcome of Aneurysmal Subarachnoid Hemorrhage Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210618
Record Dates: First submitted 2021-06-21; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-06

CONDITIONS: Optimal Cerebral Perfusion Pressure on the Outcome of aSAH Patients
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control group (No Intervention)
- Optimal MAP group (Experimental)
  Interventions: Device: Near-infrared spectroscopy (NIRS) and ICM+

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) and ICM+ — The intervention group will be given continuous NIRS and invasive blood pressure monitoring at same time. The correlation curve between the brain oxygenation index or the brain hemoglobin index (ORI/THx) and the blood pressure will be obtained through continuous monitoring. According to the correlation curve, the optimal blood pressure will be determined which provides the optimal CPP. Then the goal of blood pressure (within 5 mmHg of CPPopt) will be maintained as the target of blood pressure management for the intervention group during ICU stay.
  Arms: Optimal MAP group

SUMMARY:
Objectives: To investigate the impact of NIRS directed optimal cerebral perfusion pressure on the outcome of aSAH patients.

Study design: A multicenter, single-blinded, randomized controlled trial. Setting: Departments of critical care medicine of tertiary hospitals in China. Patients: 150 aSAH patients (≥ 18 years old) who admitted to ICU (predicted ICU duration time ≥ 24 hours)

Intervention:

Patients with aSAH will be randomly divided into the control group and the intervention group. The control group will follow the SAH guidelines. The intervention group will be given continuous NIRS and invasive blood pressure monitoring at same time. The correlation curve between the brain oxygenation index or the brain hemoglobin index (ORI/THx) and the blood pressure will be obtained through continuous monitoring. According to the correlation curve, the optimal blood pressure will be determined which provides the optimal CPP. Then the goal of blood pressure (within 5 mmHg of CPPopt) will be maintained as the target of blood pressure management for the intervention group during ICU stay.

Primary outcome: Neurological prognosis (GCS score，GOS score, and NIHSS score when discharge from ICU; GOS score at 6 months), etc.

Predicted duration of the study: 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Admitted to ICU because of aSAH.
* Predicted to stay in ICU ≥ 24 hours
* Provide written informed consent.

Exclusion Criteria:

* Unable to perform NIRS monitoring because of anatomic factors;
* Patients with severe organ failure;
* In addition to aneurysmal subarachnoid hemorrhage, there are other serious intracranial diseases (intracranial infection, cerebral hemorrhage, cerebral infarction, brain trauma, other patients after intracranial surgery);
* Patients with carotid plaque or thrombus;
* Patients with severe intracranial pneumatosis after craniotomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurological prognosis at the discharge from ICU and at 6 months | 6 months
  GOS score at 6 months

IPD SHARING:
Plan to Share IPD: Undecided